CLINICAL TRIAL: NCT00766233
Title: Phase III Study for Analysis of the Optimal Application Dose of Superficial Hyperthermia
Brief Title: Optimal Application Dose of Superficial Hyperthermia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universitätsmedizin Mannheim (Other)
Responsible Party: Principal Investigator, Frederik Wenz, Prof. Dr. med. Wenz, Universitätsmedizin Mannheim
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MA HT-PR 01
Record Dates: First submitted 2008-10-02; First posted 2008-10-03 (Estimated); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Tumors
Keywords: Hyperthermia; superficial tumor treatment; superficial tumors
MeSH Terms: conditions — Neoplasms; Hyperthermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Hyperthermal treatment once per week
  Interventions: Other: Hyperthermal treatment
- 2 (Active Comparator): Hyperthermal treatment 3 times a week
  Interventions: Other: Hyperthermal treatment

INTERVENTIONS:
Other: Hyperthermal treatment — Hyperthermal treatment one or three times per week for 60 minutes

SUMMARY:
Hyperthermia - a warming of the tumor at 42-43 ° C - in combination with radiation and / or chemotherapy is a proven method of treatment for malignant tumors. The amplification of the effect of radiotherapy and various chemotherapeutic agents (platinum analogues, nitrogen-Lost derivatives, cytotoxic antibiotics) is experimentally demonstrated. Randomized clinical trials have shown a better chance of survival and better local tumor control without increasing the toxicity of combined treatment especially also in children's tumors. The combination of hyperthermia and radiation therapy is more effective than radiotherapy alone. Hyperthermal temperatures increase blood circulation in tumors as a response to stimulation with heat. Tumor tissue, having a minor circulation and being acidotic, is resistant to radiotherapy, but sensitive to hyperthermia, while tumor with a high blood flow is sensitivity to radiation. This positive interaction is a compelling reason for the combination of hyperthermia and ionized radiation.

Hyperthermia, in combination with chemotherapy, increases the concentration of cytostatics in the tumor region, raising blood flow caused by warmth. In addition, hyperthermia increases toxicity of drugs in cells, being normally resistant to many drugs. Hyperthermia can synergistically be combined with chemotherapy treating "high risk" - tumors with curative intention.

In addition to the clinical use of surface hyperthermia (BSD 500 - O), with appropriate treatment of tumors up to 3 cm deep from the surface of the body with established indications and palliative indication in advanced stages of cancer, a prospective, randomized study with quality-controlled thermometry shall establish the optimal sequence of Hyperthermia in combination with irradiation. Therefore the treatment sequence of once per weeks is compared to a sequence of three times per week.

ELIGIBILITY:
Inclusion Criteria:

* Surficial tumors (< 3-4 cm)
* ≥ 18 years
* Karnofsky Index > 60
* No other treatment in between 30 d, applicable radiation dose min.30 Gy
* Cumulative equivalent minutes 42°C T75

Exclusion Criteria:

* Pregnancy
* Pace maker
* Metal implants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2008-01; Primary Completion 2016-01 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Complete remission (Imaging / clinical) | 5 years

SECONDARY OUTCOMES:
Progression-free survival, overall survival, Quality of life | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Radiotherapy University Hospital Mannheim, Mannheim, Germany